CLINICAL TRIAL: NCT07303790
Title: An Early Exploratory Study to Assess the Tolerability and Safety of GC012F in Patients With Multiple Sclerosis
Brief Title: This is an Early Exploratory Study to Assess the Tolerability and Safety of GC012F in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daishi Tian (Other)
Responsible Party: Sponsor-Investigator, Daishi Tian, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D831DN00001
Record Dates: First submitted 2025-12-09; First posted 2025-12-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; CAR-T cell therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: In this study, a single dose group is planned for the CAR-T cell infusion dose.Among them, 6 subjects will be enrolled in the DLT observation phase, and 9 subjects will be enrolled in the expansion phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F CAR-T Cell Injection (Experimental): This study is an early exploratory. The main purpose is an IIT clinical trial to evaluate the safety and efficacy of GC012F dual CAR-T injection in Multiple Sclerosis patinents . The enrolled patients were patients with Multiple Sclerosis .
  Interventions: Drug: GC012F CAR-T Cell Injection

INTERVENTIONS:
Drug: GC012F CAR-T Cell Injection — A single dose group is planned for the CAR-T cell infusion dose is administrated for each subject.Single IV infusion.

SUMMARY:
This is an early exploratory study to assess the tolerability and safety of GC012F CAR T cell injection in Multiple Sclerosis patients.

DETAILED DESCRIPTION:
This is a single-arm, open-label, early exploratory clinical study to evaluate the safety and efficacy of GC012F Injection in patients with MS, as well as to assess its PK and PD profiles.

This study consists of the following periods: screening period, apheresis day, baseline period, lymphodepletion preconditioning period, GC012F infusion, safety and efficacy follow-up period, and long-term follow-up period.

In this study, a single dose group is planned for the CAR-T cell infusion dose,and 15 evaluable subjects will be included. Eligible subjects will receive a single infusion of GC012F Injection and will be monitored for DLTs within 28 days following the infusion of GC012F Injection.

After all the 6 subjects have completed DLT observation, all clinical study safety data collected during the DLT observation phase will be assessed. 9 subjects will be enrolled in the dose expansion phase.

After CAR-T cell infusion, subjects will be followed up for safety, cell proliferation and survival, and efficacy until 672 days (96 weeks) after infusion, withdrawal from the study, death, withdrawal of informed consent, or lost to follow-up, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1. The laboratory test results at screening must meet the following criteria:

  * a)Absolute neutrophil count ≥ 1.0 × 10^9/L (no growth factor is given for supportive care within 7 days prior to testing);
  * b)Absolute lymphocyte count ≥ 1.0×10^9/L;
  * c)Hemoglobin ≥ 80 g/L (no red blood cell transfusion is given within 7 days prior to testing);
  * d)Platelet count ≥ 50×10^9/L (no blood transfusion is given within 7 days prior to testing);
  * e)Serum IgG ≥ 500 mg/dL;
  * f)Activated partial thromboplastin time ≤ 1.5 × upper limit of normal (ULN), prothrombin time (PT) ≤ 1.5 × ULN;
  * g)Adequate renal, hepatic, cardiopulmonary function : i.Serum alanine aminotransferase and aspartate aminotransferase ≤ 3 × ULN; ii.Total bilirubin < 2 × ULN (direct bilirubin ≤ 1.5 × ULN for subjects with Gilbert's syndrome); iii.Creatinine ≤ 2 mg/dL or creatinine clearance ≥ 60 mL/min (estimated according to the Cockcroft Gault formula); iv.Subjects with left ventricular ejection fraction ≥ 45% (performed within 8 weeks prior to apheresis) as diagnosed by echocardiography (ECHO) or multi-gated acquisition scan and no evidence of pericardial effusion as determined by ECHO and no clinically significant electrocardiographic findings; v.Baseline oxygen saturation > 92% under indoor air conditions; vi.Estimated glomerular filtration rate ≥ 60 mL/min/1.73 m^2.
* 2.Confirmed diagnosis of MS based on the 2017 McDonald diagnostic criteria and diagnosis of relapsing or progressive MS based on the 2013 Lublin phenotype criteria for multiple sclerosis;

  * Relapsing-remitting multiple sclerosis (RRMS):

    1. patients with RRMS who have failed ≥ 1 highly effective disease modifying therapy (DMT) (fingolimod, siponimod, ozanimod, and anti-leukocyte cluster of differentiation [CD] 20 monoclonal antibody therapy, etc.) (defined as at least 12 months of continuous use).
    2. At least 2 clinical relapses in the past 2 years, or 1 clinical relapse in the past 2 years with ≥ 1 new Gd-enhancing lesion on MRI, or ≥ 1 new Gd-enhancing lesion on MRI within the past 6 months; c) ≥ 2 Gd-enhancing lesions on T1-weighted brain MRI at screening.
  * Primary progressive multiple sclerosis (PPMS):

    1. patients with primary progressive MS who have failed highly effective DMT and whose disease activity has worsened recently (i.e., within 1 year) (EDSS disease progression score ≥ 0.5);
    2. no Gd-enhancing lesions on brain MRI at screening.
  * Secondary progressive multiple sclerosis (SPMS):

    1. patients with secondary progressive MS who have failed highly effective DMT and whose disease activity has worsened recently (i.e., within 1 year) (EDSS disease progression score ≥ 0.5);
    2. no Gd-enhancing lesions on brain MRI at screening.
* 3.EDSS score ≥ 2.0 and ≤ 6.5;
* 4.Documented history or confirmation at screening of the presence of oligoclonal bands or an elevated IgG index in CSF.

Exclusion Criteria:

* 1.Fungal, bacterial, viral, or other infection not controlled and/or requiring hospitalization or intravenous antimicrobial therapy within 4 weeks prior to screening. Uncomplicated urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to current therapy;
* 2.Active tuberculosis or latent tuberculosis that has not been treated appropriately prior to screening;
* 3.History of severe hypersensitivity or allergy;
* 4.Primary immunodeficiency;
* 5.Impaired cardiac function or clinically significant cardiac disease;
* 6.History of serious respiratory diseases or current serious respiratory diseases, including moderate or severe or above asthma or chronic obstructive pulmonary disease, interstitial lung disease, or pulmonary fibrosis;
* 7.Current or history of cirrhosis;
* 8.History of Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus within the past 2 years, and the need for continuous use of systemic immunosuppressants/systemic disease-modifying drugs;
* 9.Any active malignancy or history of malignancy within 5 years prior to screening. The following are exceptions: early-stage tumors that have undergone radical treatment (carcinoma in situ or stage I tumors, non-ulcerative primary melanoma with a depth < 1 mm and no lymph node involvement), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, thyroid carcinoma in situ or early-stage thyroid cancer that has undergone radical treatment, cervical carcinoma in situ, or breast cancer in situ that has undergone potentially radical treatment;
* 10.Those who have clinically significant bleeding symptoms or definite haemorrhagic diathesis within 6 months prior to screening;
* 11.Arterial or venous thrombotic events such as cerebrovascular disorders (including cerebral hemorrhage, cerebral infarction, etc), deep venous thrombosis, and/or pulmonary embolism within 6 months prior to screening;
* 12.Hematologic disorders: History of cytopenia consistent with myelodysplastic syndrome; history of sickle-cell anemia or other hemoglobinopathies;
* 13.Severe underlying medical conditions, such as:

  1. Significant clinical evidence of dementia or mental status changes;
  2. History of any other central nervous system (CNS) disorders or neurodegenerative diseases, such as epilepsy, seizure, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, and psychosis;
  3. Mental disorders or psychosocial conditions that place patients at unacceptable risk.
* 14.Positive results in any of the following tests:

  1. Positive for human immunodeficiency virus (HIV) antibody;
  2. Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) with hepatitis B virus deoxyribonucleic acid (DNA) above the lower limit of detection of the assay;
  3. Positive for hepatitis C virus (HCV) antibody with HCV ribonucleic acid (RNA) above the lower limit of detection of the assay;
  4. Positive for antibodies against human T-cell lymphotropic virus types I and II;
  5. Positive for syphilis antibody. As the immunosuppression included in this study may pose an unacceptable risk, those with active HIV infection, hepatitis B (positive for HBsAg), or HCV infection (positive for anti-HCV antibodies) are excluded. Subjects are allowed to have a previous history of hepatitis B or C, provided that viral load is shown to be below the limit of detection by quantitative polymerase chain reaction and/or nucleic acid testing. Hepatitis B surface antibodies produced following hepatitis B vaccination are not considered evidence of prior infection.
* 15.Administration of a live attenuated vaccine within 4 weeks prior to apheresis;
* 16.Receipt of a different investigational drug in a clinical trial within 4 weeks prior to apheresis, or the time interval from the last dose of the investigational drug in the previous drug clinical trial to the informed consent form (ICF) signing date is still within 5 half-lives of that drug (whichever is longer);
* 17.Splenectomy within 12 months prior to the signing of ICF;
* 18.Prior therapy targeting CD19 and/or BCMA, or CAR T product therapy against any target;
* 19.Receipt of rituximab within 6 months or ofatumumab within 4 months prior to apheresis;
* 20.Patients treated with siponimod and ozanimod within 1 month prior to apheresis;
* 21.Patients treated with fingolimod within 6 weeks prior to apheresis;
* 22.Patients treated with teriflunomide within 3 months prior to apheresis;
* 23.Major surgery within 8 weeks before the signing of ICF or planned surgery during the study (except for subjects scheduled for surgery under local anesthesia, provided that the surgery will not be performed within 2 weeks after infusion);
* 24.Previous history of organ transplantation;
* 25.Confirmed diagnosis of monophasic disease, radiologically isolated syndrome, clinically isolated syndrome, and progressive isolated sclerosis based on the 2017 McDonald criteria;
* 26.History of neuromyelitis optica spectrum disorder or myelin oligodendrocyte glycoprotein antibody-related disease, or neurological diseases suspected of MS at screening;
* 27.History of CNS or spinal cord tumors, metabolic or infectious spinal cord lesions, hereditary progressive CNS diseases, sarcoidosis, or non-MS progressive neurological diseases that interfere with study assessments;
* 28.CNS disorders, such as cerebrovascular ischemia/hemorrhage, dementia, previous or current spinal cord lesions, cerebellar diseases unrelated to MS, or other diseases deemed by the investigator to potentially interfere with neurotoxicity assessment;
* 29.History of seizures, even if seizures have been well controlled with antiepileptic drugs;
* 30.MS lesions or symptoms that have the potential to increase the risk of neurotoxicity, including but not limited to tumor-like lesions (≥ 3 cm in diameter within 5 years prior to screening) or depressed level of consciousness, and/or the presence of active, clinically significant concomitant CNS pathological changes other than MS, which may impact interpretation of study results or complicate identification or assessment of neurotoxicity;
* 31. Any contraindications to lumbar puncture (LP), including but not limited to:

  1. Known or suspected structural abnormalities of the lumbar vertebra that, in the opinion of the investigator, may interfere with the conduct of LP or increase the risk of the procedure to the subject;
  2. Risk of increased or uncontrollable bleeding, including but not limited to vascular abnormalities or tumors at or around the LP site, coagulation cascade disorders, abnormal platelet function, or abnormal platelet counts;
  3. Subjects who are taking an anticoagulant (e.g., warfarin) or an antiplatelet agent (low-dose aspirin [100 mg/day or less] is permitted) do not meet the inclusion criteria unless the investigator considers it safe for the patient to temporarily discontinue the anticoagulant or antiplatelet therapy for LP;
* 32.Subjects who are unwilling or unable to undergo MRI per protocol requirements, such as those who are unable to undergo MRI due to claustrophobia, or those with clear contraindications to MRI (e.g., metal implants, metal foreign bodies in the body, cardiac pacemakers, defibrillators, etc.);
* 33.Initiation of any DMT (except for protocol-permitted bridging therapies, such as low-dose hormones) between completion of apheresis and initiation of lymphodepletion;
* 34.Circumstances that, as judged by the investigator, may hinder the subject's full participation in the study or confuse the study results, or render participation in this study not in the subject's best interests."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) Rate | 28 days
  DLT is defined as an AE that occurs within 28 days of GC012F CAR-T product reinfusion.DLT will be evaluated according to NCI-CTCAE V5.0 criteria.
Adverse Events （AEs）Rate | Up to 15 years from treatment discontinuation
  Proportion of subjects experiencing AE within 15 years after infusion of GC012F CAR-T cell injection.

SECONDARY OUTCOMES:
GC012F T cell count in peripheral blood and cerebrospinal fluid (CSF)(Pharmacokinetic evaluation indicators) | Up to 36 months from treatment discontinuation
  Maximum observed blood and CSF concentration, time to maximum observed blood and CSF concentration, area under the bloodand CSF concentration-time curve from time zero to 28 days after infusion, last observed measurable concentration, and time to last observed measurable CAR-T cell concentration
GC012F CAR gene copy number in peripheral blood and cerebrospinal fluid (CSF)(Pharmacodynamic evaluation indicators,) | Up to 36 months from treatment discontinuation
  Observe blood and CSF the highest concentration of the CAR gene copy number
Changes in the concentration of soluble B-cell maturation antigen (BCMA) in peripheral blood | Up to 36 months from treatment discontinuation
  Observe blood the highest concentration of the BCMA
Levels of Interleukins (IL-2, IL-6, IL-8, IL-10) | Up to 84 days from treatment discontinuation
  Observe blood the highest Quantification of the cytokines Interleukins (IL-2, IL-6, IL-8, IL-10)
Iimmunoglobulins (Ig) levels in peripheral blood | Up to 15 years from treatment discontinuation
  Observe blood the highest Quantification of the immunoglobulins (Ig)
Concentration levels of neurofilament light chain protein in peripheral blood and cerebrospinal fluid (CSF) | Up to 15 years from treatment discontinuation
  Observe blood and CSF the highest concentration of neurofilament light chain protein
In kappa free light chain index levels in peripheral blood and cerebrospinal fluid CSF | Up to 36 months from treatment discontinuation
  Observe blood and CSF the highest concentration of t chain index
Percentage of subjects developing antibodies against GC012F | Up to 15 years from treatment discontinuation
  Proportion of subjects experiencing against GC012F within 15 years after infusion of GC012F CAR-T cell injection.
Annualized relapse rate in subjects with relapsing-remitting multiple sclerosis (RRMS) | Up to 15 years from treatment discontinuation
  Defined to number of MS relapses after GC012F cell infusion divided by number of years of observation
Time to first relapse | Up to 15 years from treatment discontinuation
  Defined to Time from GC012F infusion to first MS relapse
Numbers of gadolinium (Gd)-enhancing T1 lesions | Up to 15 years from treatment discontinuation
  To evaluated number of gadolinium (Gd)-enhancing T1 lesions in magnetic resonance imaging (MRI) metrics from baseline
Numbers of new or definitely enlarged T2 lesions | Up to 15 years from treatment discontinuation
  To evaluated number of new or definitely enlarged T2 lesions in magnetic resonance imaging (MRI) from baseline
Total brain volume | Up to 15 years from treatment discontinuation
  To evaluated total brain volume in magnetic resonance imaging (MRI) metrics from baseline
Numbers and volume of paramagnetic rim lesions | Up to 15 years from treatment discontinuation
  To evaluated number and volume of paramagnetic rim lesions in magnetic resonance imaging (MRI) metrics from baseline
Expanded Disability Status Scale (EDSS) grade,ranges from 0 to 10 points. | Up to 15 years from treatment discontinuation
  The expanded disability status scale (EDSS) definition is a common method used to assess neurological dysfunction in MS, based on neurological findings to determine worsening and improvement of disability. Ranges from 0 points(no neurologic impairment) to 10 points (death due to Multiple Sclerosis ), at intervals of 0.5 points.
Deep gray matter volume | Up to 15 years from treatment discontinuation discontinuation
  To evaluated deep gray matter volume in magnetic resonance imaging (MRI) metrics from baseline
Cortical volume | Up to 15 years from treatment discontinuation
  To evaluated cortical volume in magnetic resonance imaging (MRI) metrics from baseline
Levels of Interferons-γ (IFN-γ) | Up to 84 days from treatment discontinuation
  Observe blood the highest Quantification of the cytokines Interferons-γ (IFN-γ)
Levels of Tumor Necrosis Factors α (TNF-α) | Up to 84 days from treatment discontinuation
  Observe blood the highest Quantification of the cytokines Tumor Necrosis Factors α(TNF-α)

CONTACTS AND LOCATIONS:
Overall Officials: Daishi Tian, Ph.D., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science & Technology, Hubei, Hubei, China

IPD SHARING:
Plan to Share IPD: No